CLINICAL TRIAL: NCT02824809
Title: Association Between Testosterone Levels and COPD Severity Measured by BODE Index in Men
Brief Title: Association Between Testosterone Levels and COPD Severity
Acronym: COPDTESTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Asociacion Argentina Medicina Respiratoria (AAMR) (Unknown)
Responsible Party: Principal Investigator, Horacio Matias Castro, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 2413
Record Dates: First submitted 2016-07-02; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypogonadism
Keywords: hypogonadism; Chronic Obstructive Pulmonary Disease; Severity of Illness Index; Testosterone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypogonadism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The Aims of the study are estimate the association between the severity of COPD and free testosterone level and the prevalence of hypogonadism in adult men with stable COPD

ELIGIBILITY:
Inclusion Criteria:

* Adults Men ≥ 45 years
* COPD defined according to clinical diagnosis and spirometry American thoracic society ( ATS) criteria
* Stable COPD without recent acute exacerbation (less than 2 weeks)

Exclusion Criteria:

* Refusal to participate or informed consent process
* Those who are under treatment with testosterone replacement or anti-androgens
* Comorbidities: Cirrhosis, Alcoholism, cryptorchidism, panhypopituitarism, Pituitary adenoma.
* Orchiectomy
* Systemic glucocorticoids (equivalent dose ≥ 4 mg of prednisone in the last 3 weeks).
* Relative and absolute contraindications for spirometry.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with stable COPD that consult in a tertiary academic teaching hospital in Buenos Aires, Argentina
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Free testosterone Level | One day

SECONDARY OUTCOMES:
Prevalence of Hypogonadism | One day

CONTACTS AND LOCATIONS:
Overall Officials: Horacio M Castro, MD, Principal Investigator — HIBA, Buenos Aires Argentina
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided